CLINICAL TRIAL: NCT01154374
Title: A Phase II, Randomized, Controlled, Two-Center Pilot Study of the Safety and Efficacy of Topically Applied MEBO® Wound Ointment Compared to Standard of Care in Subjects With Diabetic Foot Ulcers
Brief Title: A Clinical Study of the Safety and Efficacy of MEBO® Wound Ointment in Subjects With Diabetic Foot Ulcers (Pilot)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Skingenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEBO-DFU-PILOTII-001
Record Dates: First submitted 2010-06-28; First posted 2010-06-30 (Estimated); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: Diabetic Foot Ulcers (DFUs)
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

ARMS (2):
- MEBO Wound Ointment (Experimental): Topical application twice daily
  Interventions: Drug: MEBO Wound Ointment
- Standard of Care (sterile saline moistened gauze) (Active Comparator): Topical application twice daily
  Interventions: Procedure: Standard of Care (sterile saline moistened gauze)

INTERVENTIONS:
Drug: MEBO Wound Ointment — Topical application twice daily
  Arms: MEBO Wound Ointment
Procedure: Standard of Care (sterile saline moistened gauze)
  Arms: Standard of Care (sterile saline moistened gauze)

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of MEBO in the treatment of subjects with diabetic foot ulcers (DFUs).

DETAILED DESCRIPTION:
This is a phase II, randomized, controlled, two-center pilot study designed to assess the safety and efficacy of MEBO in the treatment of subjects with DFUs. Subjects meeting entry criteria will be randomly assigned in a 1:1 ratio for up to 8 weeks of treatment with either MEBO or SOC.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥18 years of age
* Able and willing to provide informed consent
* Able and willing to comply with protocol visits and procedures
* Target ulcer duration of ≥4 weeks

Exclusion Criteria:

* Ulcer of a non-diabetic pathophysiology
* Known or suspected allergies to any of the components of MEBO
* Malignancy on target ulcer foot
* Non-compliance in the screening or run-in period

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
The incidence of complete healing of the target ulcer. | 8 weeks of treatment period

SECONDARY OUTCOMES:
Time required to achieve complete healing (days). | 8 weeks treatment period
Absolute and percentage change in ulcer surface area from baseline to endpoint. | 8 weeks treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Robert S Kirsner, MD, PhD, Study Chair — University of Miami
Locations (2):
- United States (2):
  - Blume Podiatry Group, P.C., New Haven, Connecticut
  - Boston University School of Medicine, Boston, Massachusetts